CLINICAL TRIAL: NCT05060107
Title: A Phase I Study Aiming to Assess Safety and Efficacy of a Single Intra-articular Injection of MSC-derived Exosomes (CelliStem®OA-sEV) in Patients With Moderate Knee Osteoarthritis (ExoOA-1)
Brief Title: Intra-articular Injection of MSC-derived Exosomes in Knee Osteoarthritis (ExoOA-1)
Acronym: ExoOA-1
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Francisco Espinoza (Other)
Responsible Party: Sponsor-Investigator, Francisco Espinoza, Medical Chieff Officer, Regenero / C4C, Universidad de los Andes, Chile
Organization: Universidad de los Andes, Chile (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C4C060921
Record Dates: First submitted 2021-09-14; First posted 2021-09-28 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group - sEVs (Experimental): Intra-articular knee injection of exosomes (3-5 x 10e11 particles) derived from allogeneic mesenchymal stromal cells. Single dose.
  Interventions: Biological: Exosomes (sEVs)

INTERVENTIONS:
Biological: Exosomes (sEVs) — Exosomes 3-5x10e11 particles/dose

SUMMARY:
The study aim to evaluate safety of exosomes (sEVs) from allogeneic mesenchymal stromal cells delivered by an intra-articular injection in the knee of patients with mild to moderate symptomatic osteoarthritis. The sEVs will be produced in a GMP-facility. We expect to enrolle 10 patients in this phase 1 trial and the follow-up will be up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic knee OA with VAS >50mm
* Knee OA Kellgren-Lawrence grade II to III
* Chondromalacia grade I to III
* Stable joint

Exclusion Criteria:

* Bilateral symptomatic knee OA
* Local infection
* Neoplasia
* Joint replacement
* Recent use of local steroids
* BMI > 30

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-10-05 (Estimated); Primary Completion 2023-04-05 (Estimated); Study Completion 2023-10-05 (Estimated)

PRIMARY OUTCOMES:
Adverse Event | 12 months
  Ocurrence of any adverse reactions within 12 months of treatment

SECONDARY OUTCOMES:
Incidence of injection-related pain according to VAS scale (0-100mm) | 1 week
  Pain measured by VAS scale after first week of treatment
Incidence of injection-related sinovitis according to effusion grading scale of knee joint | 1 week
  Synovitis measured by effusion grading scale (zero to 3+) after first week of treatment
Pain reduction | 52 weeks
  Change in VAS score after 52 weeks
Disability reduction | 52 weeks
  Change in Womac subscale related to function (C) after 52 weeks
Percentage of responders | 52 weeks
  According to OMERACT-OARSI Criteria Index Response after 52 weeks

IPD SHARING:
Plan to Share IPD: Undecided